CLINICAL TRIAL: NCT03394963
Title: Scientific Foundations for Developing and Validating Food-based Dietary Guidelines and a Healthy Eating Index for Ethiopia
Brief Title: Developing and Validating Food-based Dietary Guidelines and a Healthy Eating Index
Status: Completed | Type: Observational
Sponsor: Ethiopian Public Health Institute (Other Government)
Collaborators: Wageningen University (Other); Food and Agriculture Organization (FAO) (Unknown); International Food Policy Research Institute (Other)
Responsible Party: Principal Investigator, Tesfaye Hailu, Researcher and PhD student, Ethiopian Public Health Institute
Other Study IDs: A4NH-FP1-CoA1
Record Dates: First submitted 2017-12-08; First posted 2018-01-09 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Healthy
Keywords: Food-Based Dietary guideline; Healthy Eating Index; Healthy Diet; Protocol; Ethiopia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Food-based dietary guidelines for healthier diet — Develop and validate food-based dietary guideline and a healthy eating index

SUMMARY:
Among several factors contributing to the occurrence of undernutrition, micronutrient deficiencies, overnutrition, and chronic disease, unhealthy diet is one of the most important factors that need to be addressed to tackle the burden in low- and middle-income countries. To maintain healthy eating in a population, it is crucial to develop and implement country-specific food-based dietary guidelines as well as monitor the adherence of the population with the guidelines. The aim of this study is to generate evidence that will help the development and validation of food-based dietary guidelines and a healthy eating index for Ethiopia. The method to develop Ethiopian food-based dietary guidelines is adapted from the 2015 Dutch food-based dietary guidelines and the Dutch healthy diet index development and validation process, and the 1998 FAO/WHO preparation and use of food-based dietary guidelines. A multidisciplinary technical working will be established to develop FBDGs. The working group will identify key messages for the guidelines that can address priority diet-related public health problems in Ethiopia based on the evidence that will be generated by the PhD student from Wageningen University and Research. The evidence generation will begin by identifying top ten diet-related diseases that lead to high morbidity and mortality in 2016. The nutrition situation (nutritional status, dietary pattern, and nutrient gaps) analysis will be conducted to define the objectives of FBDGs. A systematic review will be conducted by formulating research questions to address the objectives of the FBDGs. The FBDGs will be translated for a specific population subgroup using linear mathematical programming and validated for cultural appropriateness, acceptability, consumer understanding and practicality of the messages. Focus group discussions and key informant interviews will be conducted to validate the FBDGs. The most recent Ethiopian national food consumption survey data collected in 2011 will be used to develop a healthy eating index (HEI). The selection of a healthy eating component of HEI will be done based on the FBDGs. Validation of a healthy eating index will be conducted by comparing the HEI score based on 24-hour recall with the HEI score based on food frequency questionnaire for population characteristics and association with micronutrient intake with or without adjusting for energy and anthropometric measurement. Developing short food frequency questionnaire (FFQ) that can be scored with the index for dietary counseling and public health practice as well as dietary gap assessment for policy recommendation will be part of the study. Validation of FFQ will be conducted by collecting primary data among women of reproductive age in 500 households in rural and urban areas of Ethiopia. The data will be analyzed using the latest version of STATA, SPSS, and NVIVO software. Correlations and other appropriate advanced statistical technique will be applied as needed to answer the objectives of the study. Ethical approval will be received from the medical ethical committee of Wageningen University and Research and scientific and ethical review office of Ethiopian Public Health Institute. This Ph.D. research is supported by the Food Systems for Healthier Diets flagship of the CGIAR- Agriculture for Nutrition and Health Programme coordinated by International Food Policy Research Institute. Food and Agriculture Organization (FAO) and Ethiopian Public Health Institute are collaborators of this project to develop the FBDGs.

DETAILED DESCRIPTION:
Triple burden of malnutrition (i.e. protein-energy malnutrition including micronutrient deficiency and overnutrition) is a current global problem. In 2017, 155 out of 677 million children in the world under the age of 5 years were stunted (height for age < -2 SD of the WHO Child Growth Standards median), 52 million wasted (weight for height < -2 SD of the WHO child growth standards median) and 41 million overweight (weight for height > 2 SD of the WHO child growth standards median) with 93 million children at risk of overweight. Out of 5 billion adults worldwide, nearly 2 billion are overweight (BMI > 25 kg/m2) or obese (BMI > 30 kg/m2) and one in 12 has a type -2 diabetes mellitus. The mean prevalence of adult obesity in the WHO data set was 7.5 ± 6.0% while adult overweight was much higher at 21.8 ± 10.2% and adult underweight was 13.4 ± 7.0%. The median ratio of overweight to underweight among women age 20 - 49 years was 5.8 in urban and 2.1 in rural areas of low- and middle-income countries (LMICs). Even many poor countries, countries in which underweight persists as a significant problem, had a fairly high prevalence of rural overweight. As compared to the overall Sub-Saharan Africa (SSA), urban prevalence of adult obesity and overweight were higher (12.5 ± 7.0% and 31.8 ± 12.8% respectively), child undernutrition was generally lower (30.4 ± 8.4% for stunting < -2SD from median height for age,15.5 ± 7.0% for underweight < -2SD from median weight for age and 12.0 ± 5.0% for wasting < -2SD from median weight for height) and adult underweight (BMI < 18.5 kg/m2) was also 10.5%. In addition to this, two billion people living in developing and developed countries are micronutrients deficient; they lack the vital vitamins and minerals needed to grow properly and live healthily. Iron, iodine, vitamin A, zinc, and folate separately or in combination are the priority micronutrient deficiencies for populations in most countries of the world. Micronutrient deficiencies have consequences throughout an individual's lifespan and are perpetuated across the generations. Thus, maternal and child malnutrition in low- and middle-income countries encompasses undernutrition and micronutrient deficiency, with a growing problem of overweight and obesity. The problem of triple burden of malnutrition is especially increasing in low- and middle-income countries mainly due to urbanization, fast economic growth, and changes in dietary pattern and lifestyle.

Ethiopia has a fast growing economy over the past 10 years, and a changing food environment, with declining shares of food expenditures and increased access to non-staples, processed foods, and sugary beverages. Stunting among young children has reduced from 57% in 2000, to 40% in 2014. Nevertheless, levels of stunting are still among the highest in the world and the contribution starts from underweight mothers whose birth outcome is a child with low birth weight. According to 2016 demographic and health survey report, the prevalence of stunting among under 5 children is 38%, wasting 9.9% and underweight 23.6%. The national nutrition survey conducted by Ethiopian Public Health Institute (EPHI) in 2015 also indicated that the prevalence of underweight (BMI<18.5 kg/m2) and overweight among women of reproductive age are 20% and 13% respectively. Overweight had increased by 10% between 2009 and 2015 according to the national nutrition survey results and other studies. The national micronutrient survey also showed that anemia, vitamin A, zinc, iodine, folate and vitamin B12 are public health problems among all population in Ethiopia. This indicates that, like other LMICs, Ethiopia is suffering from the triple burden of malnutrition.

The unhealthy diet is one of the most important risk factors that need to be addressed to tackle the triple burden of malnutrition in LMICs. The changes in the pattern of dietary risk factors in low- and middle-income countries is characterized by increases in the consumption of animal fat and protein, refined grains, and added sugar. In middle-income countries, from1989 to 2011, the percentage of individuals with consumption frequency of fish 5 + per week has decreased from 93% to 74%, that with consumption frequency of meat 5 + per week has increased from 25% to 51%, consumption frequency of fruits 1 + per week has increased from 48% to 94%, consumption frequency of salty snacks 1 + per week has increase from 22% to 64%, consumption frequency of sweet snacks has increased from 38% to 67%, and from 2004 to 2011, consumption frequency of poultry has increased from 86% to 96%. On the other hand, in Sub-Saharan African (SSA) countries, dietary micronutrient density index (average micronutrient density of the food supply based on 14 micronutrients: calcium, copper, iron, folate, magnesium, niacin, phosphorus, riboflavin, thiamin, vitamin A, vitamin B12, vitamin B6, vitamin C, and zinc using the 2011 global population-weighted Recommended Dietary Allowance [RDA]) has declined over the past 50 years. This indicates that there is a policy gap in terms of improving dietary quality for better health, prevention of diet-related diseases, and triple burden of malnutrition in LMICs setting. Promoting healthy eating in low- and middle-income countries can reduce the social inequality among the poor and rich, especially when it targets the disadvantaged population group. In general, healthy global diet can reduce global mortality by 6 - 10%, and greenhouse emission by 29-70%, reduce biodiversity loss and economic benefit up to 31 trillion US dollar and adoption of global dietary guidelines would result in 5.1 million avoided deaths per year [95% confidence interval (CI), 4.8-5.5 million] and 79 million years of life saved (CI, 75-83 million).

Besides this, lack of a healthy diet also contributes to the burden of diet-related diseases. Intakes of a diet low in fruits and vegetables and high in sodium are the leading dietary risks factors for non-communicable diseases (NCDs) burden in Ethiopia. Evidence from animal, clinical and epidemiological studies also showed that specific dietary patterns are associated with reduced risk of specific disease. Fruits and vegetables are associated with a reduction of the incidence of an esophagus, lung, stomach, and colorectum cancer and coronary heart diseases. In addition, by promoting a healthy diet, it is also possible to prevent different forms of malnutrition and micronutrient deficiencies.

A healthy diet means eating a variety of foods that can give the nutrients needed to maintain or improve health, feel good, and have adequate energy content. The nutrients include protein, carbohydrates, fat, water, vitamins, and minerals. To maintain healthy eating in a population, it is crucial to develop and implement country-specific food-based dietary guidelines and to enable tracking the adherence of the population to the food-based dietary guidelines.

Indications for dietary transitions are observed in several overall trends of Ethiopian eating habits such as increased energy intake, declining but still a dominant share of cereals in diets, and more purchased foods. Whether diets as a whole are changing towards healthier or unhealthier patterns, and how this differs between and within regions and population subgroups, is unclear. The increase in consumption of unhealthier components might be faster than that of healthy components as in many (187 countries) other countries of the world. In addition, Ethiopia's food production and supply are very vulnerable to climate change and variability (droughts in 2015-2016), which leads to temporal high levels of severe food insecurity and malnutrition which can easily affect the dietary pattern of the population. A national food consumption study conducted by EPHI sheds light on some major dietary gaps, including inadequate intake of vitamin A, calcium, folate and zinc. However, the heterogeneity of dietary patterns and dietary nutrient gaps concerns among the large diversity of consumers remain to be investigated and this heterogeneity currently limits efficient targeting of food-based interventions. Filling this knowledge gap was identified among the priorities of the nutrition research agenda of the country. Research could then support the development of food-based dietary guidelines for the general population above the age of 2 years.

Food-based dietary guidelines is a set of simple advisory statements that gives direction to consumers on healthy eating patterns to promote better nutrition and well-being and to address diet-related conditions. They provide advice on the type of food or food groups that need attention to promote more optimal nutrition and health outcomes for a target population in the country. The overall aim of food-based dietary guidelines is to promote overall health, contribute to the management of specific diet-related diseases and prevention of the risk factors, and to improve micronutrient deficiency and protein-energy malnutrition. Food-based dietary guidelines can be used for dietary advice regarding national food supply planning, better health status, reduced healthcare cost and improve work, growth and learning capacity for different population groups.

Food-based dietary guidelines should be specific to a given country, should be appropriate in terms of socio-demographic profile, nutritional status, health status, and dietary pattern to provide a framework for a healthy diet based on current nutrition recommendations. Country-specific food-based dietary guidelines are relevant due to foods that makeup diet are more than just a collection of nutrients. The nutrients in food interact differently when present as a food and the method of food preparation, processing, and cooking (i.e. food culture) influence the nutritional values of food. Food-based dietary guidelines should target the total diet, including all foods in daily meals and snacks, be based on food commonly consumed and all type of foods. The list of food groups used in FBDGs should be recognizable by consumers, permit the maximum flexibility in food choice to accommodate different eating tradition in a country and the description of food serving size should be in terms of commonly used household measures. Out of 58, only 7 African countries have FBDGs at the moment. Ethiopia is one of those African countries which do not have food-based dietary guidelines. In collaboration with FAO and other key local partners, Wageningen University and Research (WUR) and EPHI planned to develop food-based dietary guidelines for Ethiopian population above 2 years in the coming 4 years (until 2021).

The process for the development of the food-based dietary guidelines will have two major parts; the first part is developing the guidelines and advising how to use it at individual and HH level to improve dietary practice. To do this, establishing a national multidisciplinary technical working group composed of multiple concerned sectors such as ministry of health, ministry of agriculture and natural resources, ministry of livestock and fisheries, ministry of education, universities, research institute and development partners will be crucial to take into account different issues into consideration during the development and translation of the key messages in the FBDGs. The technical committee will agree on the key messages that have to be addressed on the FBDGs for the general population above 2 years based on evidence generated by WUR and EPHI on the wealth of foods, nutrients and health information, and other diet-related evidence and diet modeling. The general guidelines will translate into every day healthy dietary choices for specific population subgroups (women of reproductive age, school-age children, adolescent girls, adults and elderly) based on their dietary reference values. Food guide will be designed using the most commonly consumed foods in different regions of the country. In addition, dietary gap assessment will be done to see how far the FBDGs implementation can be possible in Ethiopia by comparing the current food supply with recommended healthy eating by the population. This will lead additional recommendations for policymakers and technical experts to set agriculture, trade and health target based on the demand formulated on Ethiopian food-based dietary guidelines. During the second part of the process, a healthy eating index will be developed which will be a measure of diet quality and relevant to evaluate the adherence to FBDGs. It is also relevant to determine the risk of diet-related diseases such as arthritis, diverticulitis, CVD, diabetes, common epithelial cancers, with colorectal cancer and mortality risk in Ethiopia for any future research. Therefore, the aim of this study is generating supportive evidence that will be useful for the development and validation of food-based dietary guidelines and a healthy eating index to Ethiopia.

ELIGIBILITY:
Inclusion Criteria:

* General population above 2 years of FBDGs development
* Women of reproductive age (15-49 years) for FBDGs validation
* Women of reproductive age (15-49 years) for HEI development and validation

Exclusion Criteria:

* population groups other than women of reproductive age for FBDGs validation, and HEI development and validation.

Ages: 2 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The FBDGs validation, a HEI and FFQ tools development and validation will target women of reproductive age (15-49 years), are not planning to move from the study and do not have a severe illness at the time of enrolment. Exclusion criteria will be a severe illness.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Amount of foods in gram per day from different food groups | From June 2018 - October 2021
  Country-specific food-based dietary guidelines
Healthy Eating Index | From June 2018 - October 2021
  Selection of the healthy eating components will be based on the food-based dietary guidelines developed for all Ethiopian above two years. Each component of a healthy eating index will have a minimum score of zero and maximum score between 5 to 20. The components will be scored in a way that a higher value indicates better adherence to the guidelines. The total healthy eating index score will not estimate an absolute energy intake rather it represents an intake per certain energy content. The total healthy eating index score (the sum of each components) ranges from 0 to 100, with higher scores indicating higher diet quality. The healthy eating index components will be categorized into adequacy, optimum, moderation, and ratio based on the healthier options provided in the food group of food-based dietary guidelines.
Calorie gap from different food groups | From June 2018 - October 2021
  Estimating the dietary gap in different food groups mentioned in the food based dietary guidelines by comparing with world health organization nutrient reference intake for different population group.

SECONDARY OUTCOMES:
Top 10 diseases based on total number of disability-adjusted life-years (DALYs) among all age and sex in Ethiopia | From June 2018 - October 2021
  Secondary data analysis from global burden of disease data
Top 10 diseases based on total number of death among all age and sex in Ethiopia | From June 2018 - October 2021
  Secondary data analysis from global burden of disease data
Current dietary assessment among different population group | From June 2018 - October 2021
  Secondary data analysis from the national food consumption survey. Estimate inadequate intake of nutrients (vitamin A, zinc, calcium and ...) and calories.
Trend in nutritional status: body mass index (weight in kilogram/ height in meter square) | From June 2018 - October 2021
  Nutrition trend analysis using demographic and health survey, other national nutrition and health surveys and desktop review of published journals
Height in meter | From June 2018 - October 2021
  Nutritional status trend analysis such as stunting (height for age < -2 SD of the WHO Child Growth Standards median) analysis using demographic and health survey, other national nutrition and health surveys and desktop review of published journals
Weight in kilogram | From June 2018 - October 2021
  Nutritional status trend analysis such as wasting (weight for height < -2 SD of the WHO child growth standards median) and underweight (weight for height < -2 SD of the WHO child growth standards median) using demographic and health survey, other national nutrition and health surveys and desktop review of published journals
Cultural acceptability of food-based dietary guidelines | From June 2018 - October 2021
  Qualitative study
Consumer understanding of food-based dietary guidelines | From June 2018 - October 2021
  Qualitative study
Implementation feasibility of food-based dietary guidelines | From June 2018 - October 2021
  Qualitative study

CONTACTS AND LOCATIONS:
Overall Officials: Inge D Brouwer, PhD, Study Director — Wageningen University; Edith Feskens, Prof., PhD, Study Chair — Wageningen University; Jeanne de Vries, PhD, Study Chair — Wageningen University
Locations (1):
- Ethiopian Public Health Institute, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: No
Once the protocol finalized and published, it will be shared.

REFERENCES:
- [Background] Muthuri SK, Francis CE, Wachira LJ, Leblanc AG, Sampson M, Onywera VO, Tremblay MS. Evidence of an overweight/obesity transition among school-aged children and youth in Sub-Saharan Africa: a systematic review. PLoS One. 2014 Mar 27;9(3):e92846. doi: 10.1371/journal.pone.0092846. eCollection 2014. PMID 24676350
- [Background] Ng M, Fleming T, Robinson M, Thomson B, Graetz N, Margono C, Mullany EC, Biryukov S, Abbafati C, Abera SF, Abraham JP, Abu-Rmeileh NM, Achoki T, AlBuhairan FS, Alemu ZA, Alfonso R, Ali MK, Ali R, Guzman NA, Ammar W, Anwari P, Banerjee A, Barquera S, Basu S, Bennett DA, Bhutta Z, Blore J, Cabral N, Nonato IC, Chang JC, Chowdhury R, Courville KJ, Criqui MH, Cundiff DK, Dabhadkar KC, Dandona L, Davis A, Dayama A, Dharmaratne SD, Ding EL, Durrani AM, Esteghamati A, Farzadfar F, Fay DF, Feigin VL, Flaxman A, Forouzanfar MH, Goto A, Green MA, Gupta R, Hafezi-Nejad N, Hankey GJ, Harewood HC, Havmoeller R, Hay S, Hernandez L, Husseini A, Idrisov BT, Ikeda N, Islami F, Jahangir E, Jassal SK, Jee SH, Jeffreys M, Jonas JB, Kabagambe EK, Khalifa SE, Kengne AP, Khader YS, Khang YH, Kim D, Kimokoti RW, Kinge JM, Kokubo Y, Kosen S, Kwan G, Lai T, Leinsalu M, Li Y, Liang X, Liu S, Logroscino G, Lotufo PA, Lu Y, Ma J, Mainoo NK, Mensah GA, Merriman TR, Mokdad AH, Moschandreas J, Naghavi M, Naheed A, Nand D, Narayan KM, Nelson EL, Neuhouser ML, Nisar MI, Ohkubo T, Oti SO, Pedroza A, Prabhakaran D, Roy N, Sampson U, Seo H, Sepanlou SG, Shibuya K, Shiri R, Shiue I, Singh GM, Singh JA, Skirbekk V, Stapelberg NJ, Sturua L, Sykes BL, Tobias M, Tran BX, Trasande L, Toyoshima H, van de Vijver S, Vasankari TJ, Veerman JL, Velasquez-Melendez G, Vlassov VV, Vollset SE, Vos T, Wang C, Wang X, Weiderpass E, Werdecker A, Wright JL, Yang YC, Yatsuya H, Yoon J, Yoon SJ, Zhao Y, Zhou M, Zhu S, Lopez AD, Murray CJ, Gakidou E. Global, regional, and national prevalence of overweight and obesity in children and adults during 1980-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2014 Aug 30;384(9945):766-81. doi: 10.1016/S0140-6736(14)60460-8. Epub 2014 May 29. PMID 24880830
- [Background] Gernand AD, Schulze KJ, Stewart CP, West KP Jr, Christian P. Micronutrient deficiencies in pregnancy worldwide: health effects and prevention. Nat Rev Endocrinol. 2016 May;12(5):274-89. doi: 10.1038/nrendo.2016.37. Epub 2016 Apr 1. PMID 27032981
- [Background] Haddad, L.J., et al., Global Nutrition Report 2015: Actions and accountability to advance nutrition and sustainable development. 2015: Intl Food Policy Res Inst.
- [Background] Tzioumis E, Adair LS. Childhood dual burden of under- and overnutrition in low- and middle-income countries: a critical review. Food Nutr Bull. 2014 Jun;35(2):230-43. doi: 10.1177/156482651403500210. PMID 25076771
- [Background] Initiatives, D., Global Nutrition Report 2017: Nourishing the SDGs. 2017.
- [Background] Mendez MA, Monteiro CA, Popkin BM. Overweight exceeds underweight among women in most developing countries. Am J Clin Nutr. 2005 Mar;81(3):714-21. doi: 10.1093/ajcn/81.3.714. PMID 15755843
- [Background] Wojcicki JM. The double burden household in sub-Saharan Africa: maternal overweight and obesity and childhood undernutrition from the year 2000: results from World Health Organization Data (WHO) and Demographic Health Surveys (DHS). BMC Public Health. 2014 Oct 31;14:1124. doi: 10.1186/1471-2458-14-1124. PMID 25361562
- [Background] Beal T, Massiot E, Arsenault JE, Smith MR, Hijmans RJ. Global trends in dietary micronutrient supplies and estimated prevalence of inadequate intakes. PLoS One. 2017 Apr 11;12(4):e0175554. doi: 10.1371/journal.pone.0175554. eCollection 2017. PMID 28399168
- [Background] Bailey RL, West KP Jr, Black RE. The epidemiology of global micronutrient deficiencies. Ann Nutr Metab. 2015;66 Suppl 2:22-33. doi: 10.1159/000371618. Epub 2015 Jun 2. PMID 26045325
- [Background] Ahmed T, Hossain M, Sanin KI. Global burden of maternal and child undernutrition and micronutrient deficiencies. Ann Nutr Metab. 2012;61 Suppl 1:8-17. doi: 10.1159/000345165. Epub 2013 Jan 21. PMID 23343943
- [Background] Nguyen PH, Gonzalez-Casanova I, Young MF, Truong TV, Hoang H, Nguyen H, Nguyen S, DiGirolamo AM, Martorell R, Ramakrishnan U. Preconception Micronutrient Supplementation with Iron and Folic Acid Compared with Folic Acid Alone Affects Linear Growth and Fine Motor Development at 2 Years of Age: A Randomized Controlled Trial in Vietnam. J Nutr. 2017 Aug;147(8):1593-1601. doi: 10.3945/jn.117.250597. Epub 2017 Jun 14. PMID 28615372
- [Background] Black RE, Victora CG, Walker SP, Bhutta ZA, Christian P, de Onis M, Ezzati M, Grantham-McGregor S, Katz J, Martorell R, Uauy R; Maternal and Child Nutrition Study Group. Maternal and child undernutrition and overweight in low-income and middle-income countries. Lancet. 2013 Aug 3;382(9890):427-451. doi: 10.1016/S0140-6736(13)60937-X. Epub 2013 Jun 6. PMID 23746772
- [Background] Popkin BM, Gordon-Larsen P. The nutrition transition: worldwide obesity dynamics and their determinants. Int J Obes Relat Metab Disord. 2004 Nov;28 Suppl 3:S2-9. doi: 10.1038/sj.ijo.0802804. PMID 15543214
- [Background] Tebekaw Y, Teller C, Colon-Ramos U. The burden of underweight and overweight among women in Addis Ababa, Ethiopia. BMC Public Health. 2014 Nov 1;14:1126. doi: 10.1186/1471-2458-14-1126. PMID 25361603
- [Background] Kimani-Murage EW, Muthuri SK, Oti SO, Mutua MK, van de Vijver S, Kyobutungi C. Evidence of a Double Burden of Malnutrition in Urban Poor Settings in Nairobi, Kenya. PLoS One. 2015 Jun 22;10(6):e0129943. doi: 10.1371/journal.pone.0129943. eCollection 2015. PMID 26098561
- [Background] Darnton-Hill I, Mkparu UC. Micronutrients in pregnancy in low- and middle-income countries. Nutrients. 2015 Mar 10;7(3):1744-68. doi: 10.3390/nu7031744. PMID 25763532
- [Background] Humphries DL, Dearden KA, Crookston BT, Woldehanna T, Penny ME, Behrman JR; Young Lives Determinants Consequences of Child Growth Project team. Household food group expenditure patterns are associated with child anthropometry at ages 5, 8 and 12 years in Ethiopia, India, Peru and Vietnam. Econ Hum Biol. 2017 Aug;26:30-41. doi: 10.1016/j.ehb.2017.02.001. Epub 2017 Feb 14. PMID 28222325
- [Background] Desalew A, Mandesh A, Semahegn A. Childhood overweight, obesity and associated factors among primary school children in dire dawa, eastern Ethiopia; a cross-sectional study. BMC Obes. 2017 Jun 1;4:20. doi: 10.1186/s40608-017-0156-2. eCollection 2017. PMID 28572983
- [Background] ICF, C.S.A.E.a., Ethiopia Demographic and Health Survey 2016: Key Indicators Report. Addis Ababa, Ethiopia, and Rockville, Maryland, USA. CSA and ICF. 2016
- [Background] EPHI, Ethiopian National Nutrition Program End-Line Survey. 2015.
- [Background] Abrha S, Shiferaw S, Ahmed KY. Overweight and obesity and its socio-demographic correlates among urban Ethiopian women: evidence from the 2011 EDHS. BMC Public Health. 2016 Jul 26;16:636. doi: 10.1186/s12889-016-3315-3. PMID 27457223
- [Background] Mr. Dilnesaw Zerfu, M.A.B., Mr. Mesert W/yohanes, Mr. Girmay Ayana, Mr. Andinet Abera, Mr Biniyam Tesfaye, Mr. Desalegn Kuche, Mr. Solomon Eshetu, Dr. Aweke Kebede, Mrs. Aregash Samuel, Mr. Temesgen Awoke, Mr. Girma Mengistu, Mr. Yosef Beyene, Mrs. Alemnesh Petros, Mr. Mekonen Sisay, Ms Tsehay Assefa, Mr. Tibebu Moges, Mr. Tesfaye Hailu, Dr.Yibeltal Assefa, Dr Amha Kebede, Ethiopian National Micronutrient Survey F.S.a.N. Research, Editor. Spetember 2016, EPHI.
- [Background] Zeba AN, Delisle HF, Renier G. Dietary patterns and physical inactivity, two contributing factors to the double burden of malnutrition among adults in Burkina Faso, West Africa. J Nutr Sci. 2014 Nov 7;3:e50. doi: 10.1017/jns.2014.11. eCollection 2014. PMID 26101618
- [Background] Fikadu T, Assegid S, Dube L. Factors associated with stunting among children of age 24 to 59 months in Meskan district, Gurage Zone, South Ethiopia: a case-control study. BMC Public Health. 2014 Aug 7;14:800. doi: 10.1186/1471-2458-14-800. PMID 25098836
- [Background] Fekadu Y, Mesfin A, Haile D, Stoecker BJ. Factors associated with nutritional status of infants and young children in Somali Region, Ethiopia: a cross- sectional study. BMC Public Health. 2015 Sep 2;15:846. doi: 10.1186/s12889-015-2190-7. PMID 26330081
- [Background] Malik VS, Willett WC, Hu FB. Global obesity: trends, risk factors and policy implications. Nat Rev Endocrinol. 2013 Jan;9(1):13-27. doi: 10.1038/nrendo.2012.199. Epub 2012 Nov 20. PMID 23165161
- [Background] Romieu I, Dossus L, Barquera S, Blottiere HM, Franks PW, Gunter M, Hwalla N, Hursting SD, Leitzmann M, Margetts B, Nishida C, Potischman N, Seidell J, Stepien M, Wang Y, Westerterp K, Winichagoon P, Wiseman M, Willett WC; IARC working group on Energy Balance and Obesity. Energy balance and obesity: what are the main drivers? Cancer Causes Control. 2017 Mar;28(3):247-258. doi: 10.1007/s10552-017-0869-z. Epub 2017 Feb 17. PMID 28210884
- [Background] Valera B, Sohani Z, Rana A, Poirier P, Anand SS. The ethnoepidemiology of obesity. Can J Cardiol. 2015 Feb;31(2):131-41. doi: 10.1016/j.cjca.2014.10.005. Epub 2014 Nov 25. PMID 25661548
- [Background] Lachat C, Otchere S, Roberfroid D, Abdulai A, Seret FM, Milesevic J, Xuereb G, Candeias V, Kolsteren P. Diet and physical activity for the prevention of noncommunicable diseases in low- and middle-income countries: a systematic policy review. PLoS Med. 2013;10(6):e1001465. doi: 10.1371/journal.pmed.1001465. Epub 2013 Jun 11. PMID 23776415
- [Background] Delobelle P, Sanders D, Puoane T, Freudenberg N. Reducing the Role of the Food, Tobacco, and Alcohol Industries in Noncommunicable Disease Risk in South Africa. Health Educ Behav. 2016 Apr;43(1 Suppl):70S-81S. doi: 10.1177/1090198115610568. PMID 27037150
- [Background] Mayen AL, de Mestral C, Zamora G, Paccaud F, Marques-Vidal P, Bovet P, Stringhini S. Interventions promoting healthy eating as a tool for reducing social inequalities in diet in low- and middle-income countries: a systematic review. Int J Equity Health. 2016 Dec 22;15(1):205. doi: 10.1186/s12939-016-0489-3. PMID 28007023
- [Background] Springmann M, Godfray HC, Rayner M, Scarborough P. Analysis and valuation of the health and climate change cobenefits of dietary change. Proc Natl Acad Sci U S A. 2016 Apr 12;113(15):4146-51. doi: 10.1073/pnas.1523119113. Epub 2016 Mar 21. PMID 27001851
- [Background] Naicker A, Venter CS, MacIntyre UE, Ellis S. Dietary quality and patterns and non-communicable disease risk of an Indian community in KwaZulu-Natal, South Africa. J Health Popul Nutr. 2015 Aug 8;33:12. doi: 10.1186/s41043-015-0013-1. PMID 26825059
- [Background] Popkin BM. Global nutrition dynamics: the world is shifting rapidly toward a diet linked with noncommunicable diseases. Am J Clin Nutr. 2006 Aug;84(2):289-98. doi: 10.1093/ajcn/84.1.289. PMID 16895874
- [Background] Melaku YA, Temesgen AM, Deribew A, Tessema GA, Deribe K, Sahle BW, Abera SF, Bekele T, Lemma F, Amare AT, Seid O, Endris K, Hiruye A, Worku A, Adams R, Taylor AW, Gill TK, Shi Z, Afshin A, Forouzanfar MH. The impact of dietary risk factors on the burden of non-communicable diseases in Ethiopia: findings from the Global Burden of Disease study 2013. Int J Behav Nutr Phys Act. 2016 Dec 16;13(1):122. doi: 10.1186/s12966-016-0447-x. PMID 27978839
- [Background] Banfield EC, Liu Y, Davis JS, Chang S, Frazier-Wood AC. Poor Adherence to US Dietary Guidelines for Children and Adolescents in the National Health and Nutrition Examination Survey Population. J Acad Nutr Diet. 2016 Jan;116(1):21-27. doi: 10.1016/j.jand.2015.08.010. Epub 2015 Sep 26. PMID 26391469
- [Background] Ptomey L, Goetz J, Lee J, Donnelly J, Sullivan D. Diet Quality of Overweight and Obese Adults with Intellectual and Developmental Disabilities as Measured by the Healthy Eating Index-2005. J Dev Phys Disabil. 2013 Dec 1;25(6):10.1007/s10882-013-9339-z. doi: 10.1007/s10882-013-9339-z. PMID 24319322
- [Background] Sekiyama M, Jiang HW, Gunawan B, Dewanti L, Honda R, Shimizu-Furusawa H, Abdoellah OS, Watanabe C. Double Burden of Malnutrition in Rural West Java: Household-Level Analysis for Father-Child and Mother-Child Pairs and the Association with Dietary Intake. Nutrients. 2015 Oct 2;7(10):8376-91. doi: 10.3390/nu7105399. PMID 26445058
- [Background] Dauchet L, Amouyel P, Hercberg S, Dallongeville J. Fruit and vegetable consumption and risk of coronary heart disease: a meta-analysis of cohort studies. J Nutr. 2006 Oct;136(10):2588-93. doi: 10.1093/jn/136.10.2588. PMID 16988131
- [Background] Riboli E, Norat T. Epidemiologic evidence of the protective effect of fruit and vegetables on cancer risk. Am J Clin Nutr. 2003 Sep;78(3 Suppl):559S-569S. doi: 10.1093/ajcn/78.3.559S. PMID 12936950
- [Background] http://www.breastcancer.org/tips/nutrition/healthy_eat. What Does Healthy Eating Mean? 2017 [cited 2017 July].
- [Background] Smitasiri S, Uauy R. Beyond recommendations: implementing food-based dietary guidelines for healthier populations. Food Nutr Bull. 2007 Mar;28(1 Suppl International):S141-51. doi: 10.1177/15648265070281S112. PMID 17521125
- [Background] Worku I, D.M., Minten B, Diet transformation in Ethiopia. 2015.
- [Background] Aurino E, Fernandes M, Penny ME. The nutrition transition and adolescents' diets in low- and middle-income countries: a cross-cohort comparison. Public Health Nutr. 2017 Jan;20(1):72-81. doi: 10.1017/S1368980016001865. Epub 2016 Jul 29. PMID 27469288
- [Background] Imamura F, Micha R, Khatibzadeh S, Fahimi S, Shi P, Powles J, Mozaffarian D; Global Burden of Diseases Nutrition and Chronic Diseases Expert Group (NutriCoDE). Dietary quality among men and women in 187 countries in 1990 and 2010: a systematic assessment. Lancet Glob Health. 2015 Mar;3(3):e132-42. doi: 10.1016/S2214-109X(14)70381-X. PMID 25701991
- [Background] Thornton PK, Ericksen PJ, Herrero M, Challinor AJ. Climate variability and vulnerability to climate change: a review. Glob Chang Biol. 2014 Nov;20(11):3313-28. doi: 10.1111/gcb.12581. Epub 2014 Apr 26. PMID 24668802
- [Background] Hagos S, Lunde T, Mariam DH, Woldehanna T, Lindtjorn B. Climate change, crop production and child under nutrition in Ethiopia; a longitudinal panel study. BMC Public Health. 2014 Aug 27;14:884. doi: 10.1186/1471-2458-14-884. PMID 25163522
- [Background] EPHI, Ethiopia National Food Consumption Survey. 2013.
- [Background] EPHI, The 2nd BSC Based EPHI's Strategic Management Plan (2015/16 to 2019/20). July 2015.
- [Background] FMOH, NATIONAL NUTRITION PROGRAM 2016-2020, Addis Ababa Ethiopia JULY 2016.
- [Background] Jankovic N, Geelen A, Streppel MT, de Groot LC, Orfanos P, van den Hooven EH, Pikhart H, Boffetta P, Trichopoulou A, Bobak M, Bueno-de-Mesquita HB, Kee F, Franco OH, Park Y, Hallmans G, Tjonneland A, May AM, Pajak A, Malyutina S, Kubinova R, Amiano P, Kampman E, Feskens EJ. Adherence to a healthy diet according to the World Health Organization guidelines and all-cause mortality in elderly adults from Europe and the United States. Am J Epidemiol. 2014 Nov 15;180(10):978-88. doi: 10.1093/aje/kwu229. Epub 2014 Oct 15. PMID 25318818
- [Background] Gibson, R.S., Principles of nutritional assessment. 2005: Oxford university press, USA.
- [Background] http://www.fao.org/nutrition/education/food-dietary-guidelines/en/. Food-based dietary guidelines. 2017 [cited 2017 July ].
- [Background] Moron C. Food-based nutrition interventions at community level. Br J Nutr. 2006 Aug;96 Suppl 1:S20-2. doi: 10.1079/bjn20061693. PMID 16923244
- [Background] Jungert A, Spinneker A, Nagel A, Neuhauser-Berthold M. Dietary intake and main food sources of vitamin D as a function of age, sex, vitamin D status, body composition, and income in an elderly German cohort. Food Nutr Res. 2014 Sep 17;58. doi: 10.3402/fnr.v58.23632. eCollection 2014. PMID 25317118
- [Background] Hunsaker SL, Jensen CD. Effectiveness of a Parent Health Report in Increasing Fruit and Vegetable Consumption Among Preschoolers and Kindergarteners. J Nutr Educ Behav. 2017 May;49(5):380-386.e1. doi: 10.1016/j.jneb.2017.01.002. Epub 2017 Feb 28. PMID 28258819
- [Background] Meegan AP, Perry IJ, Phillips CM. The Association between Dietary Quality and Dietary Guideline Adherence with Mental Health Outcomes in Adults: A Cross-Sectional Analysis. Nutrients. 2017 Mar 5;9(3):238. doi: 10.3390/nu9030238. PMID 28273871
- [Background] Brunner E, Cohen D, Toon L. Cost effectiveness of cardiovascular disease prevention strategies: a perspective on EU food based dietary guidelines. Public Health Nutr. 2001 Apr;4(2B):711-5. doi: 10.1079/phn2001161. PMID 11683566
- [Background] Bourne LT, Marais D, Love P. The process followed in the development of the paediatric food-based dietary guidelines for South Africa. Matern Child Nutr. 2007 Oct;3(4):239-50. doi: 10.1111/j.1740-8709.2007.00109.x. PMID 17824852
- [Background] Erve, I.v.t., Tulen, C. B. M., Jansen, J., Laar, A. D. E. van, Minnema, R.,Schenk, P. R., Wolvers, D., Rossum, C. T. M. van and Verhagen, H, Overview of Elements within National Food-Based Dietary Guidelines. European Journal of Nutrition & Food Safety, 2017 7(1): p. 1-56.
- [Background] Preparation and use of food-based dietary guidelines. Report of a joint FAO/WHO consultation. FAO/WHO. World Health Organ Tech Rep Ser. 1998;880:i-vi, 1-108. No abstract available. PMID 9795598
- [Background] Thorpe MG, Milte CM, Crawford D, McNaughton SA. A Revised Australian Dietary Guideline Index and Its Association with Key Sociodemographic Factors, Health Behaviors and Body Mass Index in Peri-Retirement Aged Adults. Nutrients. 2016 Mar 11;8(3):160. doi: 10.3390/nu8030160. PMID 26978399
- [Background] Acar Tek N, Yildiran H, Akbulut G, Bilici S, Koksal E, Gezmen Karadag M, Sanlier N. Evaluation of dietary quality of adolescents using Healthy Eating Index. Nutr Res Pract. 2011 Aug;5(4):322-8. doi: 10.4162/nrp.2011.5.4.322. Epub 2011 Aug 31. PMID 21994527
- [Background] Shivappa N, Hebert JR, Kivimaki M, Akbaraly T. Alternative Healthy Eating Index 2010, Dietary Inflammatory Index and risk of mortality: results from the Whitehall II cohort study and meta-analysis of previous Dietary Inflammatory Index and mortality studies. Br J Nutr. 2017 Aug;118(3):210-221. doi: 10.1017/S0007114517001908. PMID 28831955
- [Background] Kromhout D, Spaaij CJ, de Goede J, Weggemans RM. The 2015 Dutch food-based dietary guidelines. Eur J Clin Nutr. 2016 Aug;70(8):869-78. doi: 10.1038/ejcn.2016.52. Epub 2016 Apr 6. PMID 27049034
- [Background] van Lee L, Feskens EJ, Hooft van Huysduynen EJ, de Vries JH, van 't Veer P, Geelen A. The Dutch Healthy Diet index as assessed by 24 h recalls and FFQ: associations with biomarkers from a cross-sectional study. J Nutr Sci. 2014 Jan 2;2:e40. doi: 10.1017/jns.2013.28. eCollection 2013. PMID 25191596
- [Background] Looman M, Feskens EJ, de Rijk M, Meijboom S, Biesbroek S, Temme EH, de Vries J, Geelen A. Development and evaluation of the Dutch Healthy Diet index 2015. Public Health Nutr. 2017 Sep;20(13):2289-2299. doi: 10.1017/S136898001700091X. Epub 2017 Jun 19. PMID 28625202
- [Background] GBD 2016 Risk Factors Collaborators. Global, regional, and national comparative risk assessment of 84 behavioural, environmental and occupational, and metabolic risks or clusters of risks, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1345-1422. doi: 10.1016/S0140-6736(17)32366-8. PMID 28919119
- [Background] Rosner AL. Evidence-based medicine: revisiting the pyramid of priorities. J Bodyw Mov Ther. 2012 Jan;16(1):42-9. doi: 10.1016/j.jbmt.2011.05.003. Epub 2011 Jun 24. PMID 22196426
- [Background] Joint, F. and W.H. Organization, Vitamin and mineral requirements in human nutrition. 2005.
- [Background] Bowen DJ, Kreuter M, Spring B, Cofta-Woerpel L, Linnan L, Weiner D, Bakken S, Kaplan CP, Squiers L, Fabrizio C, Fernandez M. How we design feasibility studies. Am J Prev Med. 2009 May;36(5):452-7. doi: 10.1016/j.amepre.2009.02.002. PMID 19362699
- [Background] Procter-Gray E, Olendzki B, Kane K, Churchill L, Hayes RB, Aguirre A, Kang HJ, Li W. Comparison of Dietary Quality Assessment Using Food Frequency Questionnaire and 24-hour-recalls in Older Men and Women. AIMS Public Health. 2017 Jul 3;4(4):326-346. doi: 10.3934/publichealth.2017.4.326. eCollection 2017. PMID 29546221
- [Background] Mark SD, Thomas DG, Decarli A. Measurement of exposure to nutrients: an approach to the selection of informative foods. Am J Epidemiol. 1996 Mar 1;143(5):514-21. doi: 10.1093/oxfordjournals.aje.a008772. PMID 8610667
- [Background] Molag ML, de Vries JH, Ocke MC, Dagnelie PC, van den Brandt PA, Jansen MC, van Staveren WA, van't Veer P. Design characteristics of food frequency questionnaires in relation to their validity. Am J Epidemiol. 2007 Dec 15;166(12):1468-78. doi: 10.1093/aje/kwm236. Epub 2007 Sep 18. PMID 17881382
- [Background] Kuyper EM, Engle-Stone R, Arsenault JE, Arimond M, Adams KP, Dewey KG. Dietary gap assessment: an approach for evaluating whether a country's food supply can support healthy diets at the population level. Public Health Nutr. 2017 Sep;20(13):2277-2288. doi: 10.1017/S1368980017001173. Epub 2017 Jun 21. PMID 28633691
- [Derived] Bekele TH, de Vries JJ, Trijsburg L, Feskens E, Covic N, Kennedy G, Brouwer ID. Methodology for developing and evaluating food-based dietary guidelines and a Healthy Eating Index for Ethiopia: a study protocol. BMJ Open. 2019 Jul 16;9(7):e027846. doi: 10.1136/bmjopen-2018-027846. PMID 31315863